CLINICAL TRIAL: NCT05272826
Title: A Single Arm, Response-adapted, Open Label Study of Iberdomide, Weekly Bortezomib and Dexamethasone (IberBd) With Isatuximab Added on Demand for Transplant-ineligible, Newly Diagnosed Multiple Myeloma Patients: the BOREALIS Trial
Brief Title: Study of Iberdomide, Bortezomib, Dexamethasone With Isatuximab Added on Demand for ND-NTE MM Patients
Acronym: BOREALIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Myeloma Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRG 010
Record Dates: First submitted 2022-02-14; First posted 2022-03-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; Bortezomib; Dexamethasone; Calcium Dobesilate; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Iberdomide — Available as formulated capsules and administered as oral medication
  Other Names: CC-220
Drug: Bortezomib — Administered as subcutaneous injection
  Other Names: Velcade
Drug: Dexamethasone — Administered as oral medication
  Other Names: Decadron
Drug: Isatuximab — Administered as subcutaneous injection
  Other Names: Sarclisa

SUMMARY:
This study will evaluate efficacy and tolerability of iberdomide, bortezomib, dexamethasone and isatuximab on demand administered in combination for newly diagnosed transplant-ineligible multiple myeloma patients.

DETAILED DESCRIPTION:
This is a phase II, multicenter, single arm, response adapted, open label study of iberdomide, weekly bortezomib and dexamethasone (IberBd) for upfront treatment of transplant ineligible patients with Multiple Myeloma. Isatuximab will be added to treatment regimen for those who do not attain VGPR after 4 cycles of IberBd, or MRD negativity after 8 cycles of IberBd. This study will have an induction phase (cycle 1-4), an intensification phase (cycle 5-8), and a maintenance phase (cycle 9 onwards).

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign informed consent form
2. Age ≥ 65 years at the time of signing consent
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Previously untreated, transplant ineligible, symptomatic multiple myeloma as defined by the criteria below.

   Both criteria a and b must be met:
   1. Clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma
   2. Any one or more of the following myeloma defining events (MDE):

   I. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically: i.Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL) ii. Renal insufficiency: creatinine clearance 177 μmol/L (>2 mg/dL) iii. Anemia: hemoglobin value of >2 g/dL below the lower limit of normal, or a hemoglobin value <10g/dL iv. Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography-CT (PET-CT)

   II. Biomarker criteria or MDE:

   i. Clonal bone marrow plasma cell percentage ≥ 60% ii. Involved: uninvolved serum free light chain (FLC) ratio ≥100 (involved FLC level must be ≥100 mg/L) iii. > 1 focal lesions on magnetic resonance imaging (MRI) studies (at least 5 mm in size)
5. Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
6. Females of child-bearing potential (FCBP) must have a negative serum test and follow the guidelines in the pregnancy prevention program. FCBP and males must either commit to continued abstinence from heterosexual intercourse or must abide by birth control requirements as described in Appendix 9 for the pregnancy prevention program.
7. Men must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy as described in Appendix 9 of the pregnancy prevention program.
8. Life expectancy of ≥ 3 months.
9. Able to take oral medications.
10. The following laboratory results must be met within 10 days prior to first study drug administration:

    1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L. Growth factors cannot be given within 10 days of study drug administration.
    2. Serum AST and ALT ≤ 1.5 x upper limit of normal (ULN).
    3. Creatinine clearance ≥ 30 mL/min either directly measured via 24-hour urine collection or calculated using MDRD (Appendix 1).
    4. Platelet count ≥ 50 x 109/L. Platelet transfusions to help subjects meet eligibility criteria are not allowed within 10 days before study enrollment.
    5. Hemoglobin ≥ 80 g/L.

Exclusion Criteria:

1. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e. less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of treatment start]).
2. Any serious medical condition that places the patient at an unacceptable risk if he or she participates in this study. Examples of such a medical condition are, but are not limited to, patient with unstable cardiac disease as defined by: Cardiac events such as MI within the past 6 months, NYHA heart failure class III-IV, uncontrolled atrial fibrillation or hypertension; patients with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
3. Pregnant or lactating females.
4. Renal failure requiring hemodialysis or peritoneal dialysis.
5. Prior history of malignancies, other than multiple myeloma, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
6. Patients who are unable or unwilling to undergo antithrombotic therapy.
7. Peripheral neuropathy of ≥ grade 2 severity.
8. Known HIV positivity or active infectious hepatitis, type A, B, or C.
9. Primary AL (immunoglobulin light chain) amyloidosis and myeloma complicated by amyloidosis.
10. Plasma Cell Leukemia
11. Evidence of cardiovascular risk including any of the following:

    1. QTc interval ≥ 470 msecs. Note that the QT interval should be corrected for heart rate by Fridericia's formula (QTcF)
    2. Evidence of current clinically significant uncontrolled arrhythmias; including clinically significant ECG abnormalities; including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
    3. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of screening.
    4. Class III or IV heart failure as defined by the New York Heart Association functional classification system (Appendix 2)
    5. Uncontrolled hypertension
12. Patients with hypersensitivity to boron or any of its excipients or to the active substance of Iberdomide or its excipients
13. Patients requiring strong inhibitors or inducers of CYP3A4/5. See Appendix 10 for a list of these drugs
14. Any concurrent severe and/or uncontrolled medical condition or psychiatric disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study or that confounds the ability to interpret data from the study.
15. Patients that have had severe acute respiratory syndrome coronavirus 2 infection within 14 days for mild or asymptomatic infections or 28 days for severe/critical illness prior to initiating study treatment.
16. Patients that have undergone major surgery (as defined by the investigator) within 28 days of initiating study treatment.
17. Active systemic infection that is likely to interfere with the study procedures or results or that, in the opinion of the investigator, would constitute a hazard for participating in this study.
18. Patients with a gastrointestinal disease that may significantly alter the absorption of iberdomide
19. Patients that have received a live vaccine within 3 months of initiating study treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate Rate of Stringent Complete Response (sCR) transplant ineligible multiple myeloma patients. | After 4 cycles of therapy (each cycle is 28 days)
  Evaluate the rate of stringent complete response (sCR) after 4 cycles of therapy of Iber+ weekly Bd in newly diagnosed transplant ineligible multiple myeloma patients.

SECONDARY OUTCOMES:
Evaluate Objective Response | After 4 cycles of therapy (each cycle is 28 days)
  Evaluate objective response as per IMWG criteria: progressive disease, stable disease, partial response, very good partial response, complete response and stringent complete response according to IMWG criteria. Multiple measurements will be aggregated to arrive at one reported value (e.g., weight and height will be combined to report BMI in kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Martha Louzada, MD, MSc, Principal Investigator — London Health Sciences Centre
Locations (5):
- Canada (5):
  - QEII Health Science Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No